CLINICAL TRIAL: NCT00904111
Title: A Randomized, Double-blind Study Comparing The Efficacy And Safety Of Lidocaine 5% Patch With Placebo In Patients With Chronic Axial Low Back Pain
Brief Title: A Study Comparing The Efficacy And Safety Of Lidocaine 5% Patch With Placebo In Patients With Chronic Axial Low Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sr. Director, Clinical R&D, Endo Pharmaceuticals Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EN3261-001
Record Dates: First submitted 2009-05-15; First posted 2009-05-19 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2010-02

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — Lidoderm; Lidocaine; Transdermal Patch

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Lidocaine 5% Patch (Experimental): Lidocaine 5% patch (Lidoderm®,Endo Pharmaceuticals Inc.), 2 patches applied directly to the most painful area of the low back once daily (q24h)
  Interventions: Drug: Lidoderm®
- Placebo Topical Patch (Placebo Comparator): Matching placebo patch, 2 patches applied directly to the most painful area of the low back once daily (q24h)
  Interventions: Drug: Placebo Topical Patch

INTERVENTIONS:
Drug: Lidoderm® — Eligible patients were randomly allocated to receive one of two treatments for 12 weeks: lidocaine 5% patch or matching placebo patch.
  Other Names: Lidocaine 5% Patch
  Arms: Lidocaine 5% Patch
Drug: Placebo Topical Patch — Eligible patients were randomly allocated to receive one of two treatments for 12 weeks: lidocaine 5% patch or matching placebo patch.
  Arms: Placebo Topical Patch

SUMMARY:
Patients with Chronic Axial Low Back Pain participated in a Phase II clinical trial to assess the efficacy of lidocaine 5% patch compared with placebo.

ELIGIBILITY:
Key Inclusion Criteria:

* Had axial LBP with or without radiation present for at least 3 months as defined as:

  * Chronic axial LBP without radiation: pain isolated to the axial low back without radiation into the buttock or below
  * Chronic axial LBP with radiation: pain that radiates to the buttock or below. This patient group could include patients with radicular/neuropathic and non-radicular components with leg pain component <50%
* Had daily moderate to severe LBP as the primary source of pain
* Had a normal neurological examination, including:

  * Motor strength
  * Sensory exam in lower extremities
  * Deep tendon reflexes
* Had a normal 12-lead electrocardiogram (ECG) without any clinically significant abnormalities in heart rate, rhythm, or conduction
* Had discontinued use of all analgesic medications (including over-the-counter [OTC] analgesics) prior to randomization (patients were allowed limited use of analgesic medications for indications other than non-study pain).
* Had a daily average pain intensity rating of 6 or greater (on a 0 to 10 scale) for at least 3 days out of the 5 consecutive days immediately prior to the baseline visit; 0 was defined as "no pain" and 10 was defined as "pain as bad as ever imagined" as measured by Question 5 of the Brief Pain Inventory (BPI) and recorded in a diary

Key Exclusion Criteria:

* Had spinal stenosis with > 50% leg pain component
* Had elective surgery scheduled to occur during the 14-week study
* Had a history of one or more back surgeries within 1 year of study entry
* Had severe renal insufficiency (creatinine clearance of <30mL/min)
* Had moderate or greater hepatic impairment
* Were taking analgesic medications that could not be discontinued during the study. Patients taking these medications prior to the study were required to discontinue use for the duration of the study. Patients using opioid analgesics at study entry were required to taper off these medications.
* Were taking long-acting opioids or opioids that could not be discontinued over the first 5 days of the placebo run-in period
* Had received an epidural steroid/local anesthesia injection within 4 weeks prior to study entry
* Had received trigger point injections within 2 weeks prior to study entry
* Had received Botulinum Toxin (Botox) Injections for LBP within 6 months prior to study entry
* Were using a lidocaine-containing product that could not be discontinued during the study
* Were using any topical medication applied to the low back region
* Had previously failed treatment with Lidoderm analgesic patch for LBP
* Were taking class 1 anti-arrhythmic drugs (e.g. mexiletine, tocainide)
* Had any other chronic pain condition that, in the opinion of the investigator, would have interfered with patient assessment of LBP relief

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2004-08; Primary Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Pain intensity (Question 5 of the BPI) | Visit - V2 (Day 0), V3 (Day 14), V4 (Day 28), V5 (Day 42), V6 (Day56), V7/EOS (Day 84)

SECONDARY OUTCOMES:
Safety Assessments included AEs, dermal assessments, clinical laboratory results (including urinalysis), vital sign measurements, physical and neurological examinations, plasma lidocaine concentration | Visit - V2 (Day 0), V3 (Day 14), V4 (Day 28), V5 (Day 42), V6 (Day56), V7/EOS (Day 84)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Endo Pharmaceuticals
Locations (18):
- United States (18):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Carlsbad, California
  - National City, California
  - Waterbury, Connecticut
  - Washington D.C., District of Columbia
  - Port Orange, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Overland Park, Kansas
  - Pittsfield, Massachusetts
  - Burlington, North Carolina
  - Altoona, Pennsylvania
  - Duncansville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Cordova, Tennessee
  - San Antonio, Texas
  - Virginia Beach, Virginia